CLINICAL TRIAL: NCT00118170
Title: Pharmacokinetic and Phase I Study of Sorafenib (BAY 43-9006, NSC 724772, IND 69896) for Solid Tumors and Hematologic Malignancies in Patients With Hepatic or Renal Dysfunction
Brief Title: Sorafenib in Treating Patients With Metastatic or Unresectable Solid Tumors, Multiple Myeloma, or Non-Hodgkin's Lymphoma With or Without Impaired Liver or Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03083; CALGB-60301; U10CA031946 (NIH); CDR0000433342 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Multiple Myeloma; Splenic Marginal Zone Lymphoma; Stage II Multiple Myeloma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib once on day 1 and then once daily, twice daily, or every other day beginning on day 8 and continuing for 3 months. Patients are re-evaluated at 3 months. Patients with responding disease may continue study treatment in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients (per treatment cohort) receive escalating doses of sorafenib until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.
  Interventions: Drug: sorafenib tosylate; Other: pharmacological study

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of sorafenib in treating patients with metastatic or unresectable solid tumors, multiple myeloma, or non-Hodgkin's lymphoma with or without impaired liver or kidney function. Sorafenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Sorafenib may have different effects in patients who have changes in their liver or kidney function

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the pharmacokinetics of BAY 43-9006 in patients with hepatic or renal dysfunction (part 1 of the study).

II. To determine a tolerable starting dose of BAY 43-9006 in patients with varying degrees of hepatic or renal dysfunction (part 2 of the study).

OUTLINE: This is a dose-escalation, multicenter study. Patients are assigned to 1 of 9 treatment cohorts according to hepatic or renal function.

Patients receive oral sorafenib once on day 1 and then once daily, twice daily, or every other day beginning on day 8 and continuing for 3 months. Patients are re-evaluated at 3 months. Patients with responding disease may continue study treatment in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients (per treatment cohort) receive escalating doses of sorafenib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have cytologically or histologically confirmed tumors that are metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; Patients with solid tumors, multiple myeloma, or non-Hodgkin's lymphoma are eligible
* Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan
* All other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly nonmeasurable lesions; Lesions that are considered non-measurable include the following:

  * Bone lesions
  * Ascites
  * Pleural/pericardial effusion
  * Lymphangitis cutis/pulmonis
  * Abdominal masses that are not confirmed and followed by imaging techniques
  * Cystic lesions
* ≥ 4 weeks since major surgery
* ≥ 4 weeks since completion of radiation or chemotherapy except for ≥ 6 weeks for nitrosoureas, L-PAM or mitomycin-C
* ECOG Performance Status of 0-2
* Non-pregnant and non-nursing because the effects of BAY 43-9006 on the fetus/infant are unknown; in addition, women of child-bearing potential and men must agree to use an appropriate method of birth control throughout their participation in this study; appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives (Norplant), or double barrier methods (diaphragm plus condom)
* No patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, or psychiatric illness/social situations that would limit compliance with study requirements
* No concomitant medications known to cause hepatic or renal toxicity, including anti-seizure medications, non-steroidal anti-inflammatory agents, and steroids
* No gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease
* No HIV-positive patients receiving combination anti-retroviral therapy because of possible pharmacokinetic interactions with BAY 43-9006; however, patients who are HIV+ but without AIDS defining diagnosis and not on combination anti-retroviral therapy are eligible
* No patients with evidence of biliary or renal obstruction; patients should be observed for at least one week after treatment (i.e. stents or drains) for biliary or renal obstruction to ensure their organ dysfunction has stabilized before registration to this protocol
* No current treatment with other investigational agents
* No evidence of bleeding diathesis
* No patients on therapeutic anticoagulation; prophylactic anticoagulation (i.e., low dose warfarin) of venous or arterial access devices is allowed provided that the requirements for PT, INR or PTT is met
* No treatment with cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or Phenobarbital), rifampin or St. John's wort
* Patients with brain metastases are eligible if they meet all of the following criteria:

  * Asymptomatic
  * Radiographically stable disease for at least 2 months
  * Previously received treatment for the brain metastases
  * Not currently receiving steroid therapy or enzyme-inducing anticonvulsants (e.g. phenytoin, phenobarbital, or carbamazepine)
* Granulocytes ≥ 1,500/μl
* Platelet count ≥ 75,000/μl
* Normal or abnormal organ function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2004-10; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Relationship between the pharmacokinetics and measures of renal dysfunction categorized by creatinine clearance as estimated by the Cockcroft and Gault formula (Part 1) | Prior to and at 1, 2, 3, 4, 6, and 24 hours post-dose on day 1
  Explored using standard parametric and non-parametric methods for one- and two-way analysis of variance (ANOVA) layouts (the dysfunction factor (hepatic/renal) and the severity factor (mild, moderate, severe, very severe).
Severity of hepatic disease as assessed by the Child-Pugh criteria | Up to 3 months
  Non-parametric measures of association for ordinal data will be employed.
Distribution of and association patterns between the Child-Pugh score and that of patient's risk of toxicity beyond each dose or cohort, assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 | Up to 5 years
Mean levels of area under the curve (AUC) using the ANOVA model | Up to 12 weeks
  90% confidence intervals for the relative change (from mild to moderate and from moderate to severe) of the mean AUC levels will be calculated.
Maximum tolerated dose (MTD) of sorafenib tosylate, assessed using the NCI CTCAE v3.0 (Part 2) | Up to 4 weeks
Dose-limiting toxicities (DLT), defined as any grade 3 or greater non-hematologic toxicity, assessed using the NCI CTCAE v3.0 | Up to 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonius Miller, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B (CALGB) Research Base, Chicago, Illinois, United States